CLINICAL TRIAL: NCT05893030
Title: Prevention of Organ Dysfunction and Mortality by Monitoring the Administration of Opioids and Hypnotics in Patients at High Postoperative Risk: the Opti-Two Study. A Multi-center Controlled Randomized Study.
Brief Title: Prevention of Organ Dysfunction and Mortality by Monitoring the Administration of Opioids and Hypnotics in Patients at High Postoperative Risk
Acronym: OPTI-TWO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Direction Générale de l'Offre de Soins (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20PH283; ANSM (Other: 2022-A01122-41)
Record Dates: First submitted 2023-05-22; First posted 2023-06-07 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Sedation and Analgesia Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental)
  Interventions: Procedure: anesthesia guided by sedation and analgesia monitoring
- Control Group (Placebo Comparator)
  Interventions: Procedure: anesthesia performed according only to the clinical judgment of the anesthetist as usual practice

INTERVENTIONS:
Procedure: anesthesia guided by sedation and analgesia monitoring — Anesthesia guided by sedation and analgesia monitoring The level of sedation will be monitored by
  * Monitoring System BIS™ : Bispectral index (BIS) between 45 and 60 AND Suppression Ratio (SR) at 0;
  * or SedLine® Sedation Monitor : Patient State Index (PSi) between 25 and 50;
  * or Entropy Sensor™: State entropy (SE) between 45 and 60 AND Burst Suppression Ratio (BSR) at 0;
  and the level of nociception by :
  * Nociception monitor PMD-200® : Nociception Level (NoL) between 10 and 25.
  Arms: Intervention Group
Procedure: anesthesia performed according only to the clinical judgment of the anesthetist as usual practice — Administration of anesthesia will be performed according to the clinical judgment of the anesthetist as usual practice without sedation and analgesia monitoring
  Arms: Control Group

SUMMARY:
Intraoperative hypotension is a common situation. It increases postoperative morbidity and mortality, especially in patients at high postoperative risk undergoing high-risk surgery. Intraoperative hypotension is partly related to anesthesia, and mainly to the combined, dose-dependent, synergistic effect of hypnotics and opioids. Monitoring sedation and monitoring analgesia reduce intraoperative consumption of each anesthetic agent. To date, the beneficial effect of combined sedation and analgesia monitoring on the reduction of intraoperative hypotension has only been found in one study, involving major abdominal surgery. Up to now, no study has been designed to demonstrate the benefit of monitoring the two components of anesthesia on postoperative organ dysfunction and mortality.

The study propose to evaluate the relevance of a combined optimization of hypnotic and opioid agents on the most frequently encountered dysfunctions related to intraoperative hypotension.

ELIGIBILITY:
Inclusion Criteria:

* patients affiliated to the French Social Security;
* informed and signed consent to participating in the study;
* planned postoperative hospitalization > 48 hours;
* patients over 75 years of age with at least one of the following postoperative risk factors:

  * ischemic coronary disease;
  * history of compensated or prior heart failure;
  * stroke;
  * significant arrhythmias: fibrillation or auricular flutter with ventricular response > 100/minute, multiform QRS complex) or cardiac conduction abnormalities (trifascicular block, auriculoventricular block of the second or third degree);
  * peripheral vascular disease;
  * chronic obstructive pulmonary disease;
  * chronic respiratory failure;
  * renal insufficiency, defined by a creatinine > 175 µmol.l-1 (2 mg.dl-1);
  * insulin therapy for diabetes;
  * active cancer;
  * chronic alcohol abuse;
  * dementia.
* elective or emergency high-risk surgery under general anesthesia with a combination of hypnotic and opioid, and intubation or placement of a supraglottic airway control device:

Non inclusion criteria:

* Patients who meet one or more of the preoperative following criteria will not be included:
* acute heart failure or acute myocardial infarction;
* acute respiratory failure or pneumonia;
* septic shock;
* acute stroke;
* cardiac surgery;
* open chest surgery;
* opioid free anesthesia;
* intraoperative ketamine at a dose > 0.2 mg.kg-1;
* lidocaine or dexmedetomidine by continuous infusion;
* refusal to participate in the study;

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1132 (Estimated)
Dates: Start 2023-10-12 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
death | Day 30
Postoperative acute kidney injury (PO-AKI) | Day 30
  The PO-AKI will be defined as an increase to 1.5 times the reference level, or as more than 0.3 mg.dl-1 (i.e. 26.5 µmol.l-1) between the last preoperative value and the maximal value observed after surgery, or urine volume < 0.5 ml.kg-1.h-1 for 6 hours, according to the recommendations of the Acute Kidney Injury Network
cardiovascular complication | Day 30
  postoperative myocardial infarction, acute heart failure, acute/non pre-existing atrial fibrillation or flutter, cardiac arrest with successful resuscitation, coronary revascularisation
neurological complication | Day 30
  Stroke or transient ischemic attack
Post-operative delirium (POD) | Day 30
  Post-operative delirium (POD) will be evaluated using the 3-minute Diagnostic Confusion Assessment Method (3D-CAM), appropriated and validated for the assessment of delirium in the postoperative period, or the Confusion Assessment Method for Intensive Care Unit (CAM-ICU) for the intubated patients.

SECONDARY OUTCOMES:
doses of hypnotics administered | during surgery
doses opioids administered; | during surgery
number and duration of hypotensive periods | during surgery
  an hypotensive event will be defined as a Mean Arterial Pressure (MAP) ≤ 65 mmHg.
time spent within the desired range of sedation: | during surgery
  Monitoring System BIS™ : Bispectral index (BIS) between 45 and 60 AND Suppression Ratio (SR) at 0 or SedLine® Sedation Monitor : Patient State Index (PSI) between 25 and 50 AND Suppression Ratio (SR) at 0 or Entropy Sensor™: State entropy (SE) between 45 and 60 AND Burst Suppression Ratio (BSR) at 0 The anesthetist will have access to the value of sedation monitoring in the "intervention" group; these data will be recorded but not available to the anesthetist in the "control" group: they will be analyzed at the end of the study to answer this point.
time spent within the desired range of analgesia: | during surgery
  Nociception monitor PMD-200® : Nociception Level (NOL) between 10 and 25. The anesthetist will have access to the value of sedation and analgesia monitoring in the "intervention" group; these data will be recorded but not available to the anesthetist in the "control" group: they will be analyzed at the end of the study to answer this point.
doses of vasopressive amines (ephedrine or norepinephrine) administered; | during surgery
pain ≥ 5 as assessed with the Visual Analogic Scale (VAS) | At 48 Hours after surgery
  VAS 0 to 10 [0 corresponds to no pain - 10 corresponds to maximum pain]
dose of opioid administered; | At 48 Hours after surgery
incidence of awareness and recall during anesthesia (explicit memory). | At 48 Hours after surgery
acute respiratory failure or Acute Respiratory Distress Syndrome (ARDS) | Day 30
duration of stay in Intensive Care Unit (ICU); | Day 30
rate of unexpected ICU admission, or readmission | Day 30
duration of hospital stay; | Day 30
early hospital readmission rate | Day 30

CONTACTS AND LOCATIONS:
Overall Officials: David CHARIER, MD, Principal Investigator — CHU DE SAINT-ETIENNE
Locations (14):
- France (14):
  - Chu D'Amiens Picardie, Amiens
  - Chru de Besancon, Besançon
  - Chu Clermont-Ferrand, Clermont-Ferrand
  - Chu de Grenoble, Grenoble
  - Chu de Lille, Lille
  - APHM - Centre Hôpital Marseille Nord, Marseille
  - Chu de Nantes, Nantes
  - Chu de Nimes, Nîmes
  - Hopital Bichat Claude Bernard, Paris
  - Chu Lyon Sud, Pierre-Bénite
  - Chu de Poitiers, Poitiers
  - Chu St-Etienne, Saint-Etienne
  - Chu de Toulouse, Toulouse
  - Médipole Lyon Villeurbanne, Villeurbanne

IPD SHARING:
Plan to Share IPD: No